CLINICAL TRIAL: NCT02978755
Title: Open, Non Controlled, Multicenter, First-in-Human Study for the Evaluation of the Safety, Pharmacokinetics and Preliminary Antitumor Activity of GM102 in Patients With Advanced Pretreated Gynecological Cancer
Brief Title: First In Human Safety, Pharmacokinetics and Anti-tumoral Activity of GM102 in Gynecological Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GamaMabs Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C101
Record Dates: First submitted 2016-11-23; First posted 2016-12-01 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Neoplasm, Gynecologic
MeSH Terms: conditions — Genital Neoplasms, Female

STUDY DESIGN:
Intervention Model Description: * phase 1 escalation GM102 single agent
  * phase 1 escalation GM102 combined with paclitaxel and carboplatin
  * phase 1b: 3 parallel expansion cohorts at the recommended dose of GM102 single agent
Oversight: Data Monitoring Committee: No

ARMS (3):
- GM102 escalating doses (Experimental): 8 successive cohorts
  Interventions: Drug: GM102
- GM102 escalating doses + carboplatin+paclitaxel (Experimental): 2 successive cohorts
  Interventions: Drug: GM102 escalating doses
- GM102 recommended dose (Experimental): 3 parallel cohorts in sex cord stromal, epithelial ovarian and cervix cancers
  Interventions: Drug: GM102

INTERVENTIONS:
Drug: GM102 — GM102 escalating doses (phase1)
  Arms: GM102 escalating doses
Drug: GM102 escalating doses — GM102 escalating doses combined with paclitaxel and carboplatin
  Arms: GM102 escalating doses + carboplatin+paclitaxel
Drug: GM102 — GM102 single agent at recommended dose in 3 parallel cohorts (sex cord, epithelial ovarian, cervix cancers)
  Arms: GM102 recommended dose

SUMMARY:
First in Human study, assessing the safety profile, the pharmacokinetics and preliminary antitumor activity of GM102, a new compound (a monoclonal antibody), in patients with previously treated gynecological cancers bearing the AMHRII (anti-mullerian Hormone Receptor II) receptor. The primary objective of the study is to determine the GM102 recommended dose.

DETAILED DESCRIPTION:
AMHRII, an embryonic receptor, is reexpressed in a subset of gynecological cancers. GM102 is a humanized low fucose monoclonal antibody with a high affinity to AMHRII receptor. GM102 acts through enhanced capability to engage immune effector cells (macrophages, natural killer (NK) cells) to trigger ADCC (antibody dependent cellular cytotoxicity) and phagocytosis of tumor cells.

Patients with gynecological tumors expressing AMHRII receptor on the tumor cells in archived tissue as determined prior to study entry will be eligible for C101 study.

C101 consists in a phase I part (dose and schedule escalation) and a phase Ib part (expansion).

The phase I part is designed to determine the recommended phase 2 dose (RP2D) using the classical 3+3 dose-finding design. In six successive escalating dose cohorts, patients will receive GM102 infusions every 2 weeks until progression or toxicity. In 4 additional cohorts, patients will receive GM102 infusions weekly until progression or toxicity and GM102 infusions combined with chemotherapy until progression or toxicity.

A Trial Steering Committee (TSC) will analyze and qualify the toxicities and will provide recommendations according to the dose administration rules defined in the protocol.

At the end of the phase I part, the RP2D will be determined, taking into account dose limiting toxicities (DLTs), overall toxicity, pharmacokinetics and pharmacodynamic effects of GM102.

The Phase Ib part of the study will confirm the tolerance of the selected dose (RP2D) and will assess antitumoral activity of GM102 in three parallel cohorts of patients with Sex Cord-Stromal tumors, and AMHRII positive ovarian and cervix cancers. Patients will be treated until progression or toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, or metastatic recurrent gynecological cancer, for whom no standard alternative therapy is available, having received at least one line of therapy and expressing AMHRII on tumor cells.
* If possible at least one lesion should be identified for 2 biopsies: a baseline biopsy and an under-treatment biopsy for AMHRII expression and GM102 pharmacodynamics evaluation.
* Available tumor block or at least 10 slides from formalin-fixed paraffin-embedded (FFPE) archival tissue.
* At least one measurable lesion by RECIST (Response Evaluation Criteria in Solid Tumors) on screening CT-scan.
* Written Informed Consent forms.
* Willing and able to comply with the trial requirements.
* Covered by healthcare insurance in accordance with local requirements.

For phase 1b, only patients with either Sex cord stromal tumors or epithelial ovarian cancer or cervix cancer will be eligible

Exclusion Criteria:

* Age < 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status > 1
* Life expectancy < 12 weeks.
* Known or symptomatic brain metastasis (other than totally resected or previously irradiated and non-progressive/relapsing) or lepto-meningeal carcinomatosis.
* Concurrent treatment with any other anticancer therapy.
* Concurrent chronic corticosteroid treatment.
* Known severe anaphylactic or other hypersensitivity reactions secondary to a prior exposure to human antibodies or to any protein product.
* Washout period before treatment initiation: < 3 weeks or 5 times the half-life, whichever is shorter, for prior antitumor therapy (small molecules and/or antibody-drug conjugates, radiotherapy) or 6 weeks for monoclonal antibodies.
* Any active concomitant malignancy.
* Serious concomitant illness e.g. active infection requiring systemic antibiotic, antifungal or antiviral drug, or physical examination or laboratory abnormalities, that, in the opinion of the Investigator, would compromise protocol objectives.
* Poor bone marrow reserve as defined by neutrophils < 1.0 x 10E9/L or haemoglobin < 9.0 g/dL or platelet count < 100 x 10E9/L.
* Poor organ function as defined by any one of the following: left ventricular ejection fraction ≤ 40%, serum creatinine > 1.5 x upper limit of normal (ULN), total bilirubin > 1.5 x ULN, AST and ALT> 2.5 x ULN in the absence of liver metastasis or > 5 x ULN in case of documented liver metastasis.
* Non-resolution of any prior treatment related toxicity to < Grade 2, except for alopecia according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03.
* Pregnancy or breastfeeding.
* Patient with reproductive potential who do not agree to use an accepted effective method of contraception - investigator's judgment - during the study period and for at least 4 months following completion of study treatment.
* Patient participating in another clinical trial investigating a treatment during the study and within 30 days prior to first study treatment administration.
* Patient deprived of her liberty by a judicial or administrative decision, patient admitted to a hospital, social institution or who is under a measure of legal protection, patient hospitalized without consent or who is in an emergency situation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-06; Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Phase I part: incidence of Dose Limiting Toxicities (DLTs) | Four weeks
  Number of patients in the DLT evaluable population experiencing at least one DLT
Phase Ib part: incidence of Serious Adverse Events (SAEs) and Treatment-Emergent Adverse Events (TEAEs) at Recommended Phase 2 Dose (RP2D) | Through study completion, an average of 1 year
  Number of patients with at least one AE

SECONDARY OUTCOMES:
PK: Maximum Serum Concentration [Cmax] | up to 16 weeks
  Cycle 1 Day 1 pre-dose, Cycle 1 Day 1 End Of Infusion (EOI), Cycle 1 Day 1 EOI + 3 hours, Cycle 1 Day 2, Cycle 1 Day 3, Cycle 1 Day 8, Cycle 1 Day 15 pre-dose, Cycle 1 Day 15 EOI, Cycle 2 Day 1 pre-dose, Cycle 2 Day 1 EOI, Cycle 2 Day 15 pre-dose, Cycle 2 Day 15 EOI, Cycle 3 Day 1 pre-dose, Cycle 3 Day 1 EOI, Cycle 3 Day 15 pre-dose, Cycle 3 Day 15 EOI, Cycle 4 Day 1 pre-dose, Cycle 4 Day 1 EOI, Cycle 4 Day 15 pre-dose, Cycle 4 Day 15 EOI
PK: Area Under the Curve [AUC] | up to 16 weeks
  Cycle 1 Day 1 pre-dose, Cycle 1 Day 1 End Of Infusion (EOI), Cycle 1 Day 1 EOI + 3 hours, Cycle 1 Day 2, Cycle 1 Day 3, Cycle 1 Day 8, Cycle 1 Day 15 pre-dose, Cycle 1 Day 15 EOI, Cycle 2 Day 1 pre-dose, Cycle 2 Day 1 EOI, Cycle 2 Day 15 pre-dose, Cycle 2 Day 15 EOI, Cycle 3 Day 1 pre-dose, Cycle 3 Day 1 EOI, Cycle 3 Day 15 pre-dose, Cycle 3 Day 15 EOI, Cycle 4 Day 1 pre-dose, Cycle 4 Day 1 EOI, Cycle 4 Day 15 pre-dose, Cycle 4 Day 15 EOI
Response Rate using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | Through study completion
  Percentage of patients who achieved a Complete Response (CR) or a Partial Response (PR) based on RECIST version 1.1
Clinical benefit rate | up to 3 months
  Percentage of patients achieving Complete Response (CR), Partial Response (PR) or Stable Disease (SD) superior to 3 months
Duration of response | Through study completion
  Duration of overall response in months for patients who achieved PR and/or CR
Time to progression (TTP) | Through study completion
  Time from first dose received until objective tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Leary, MD/PhD, Principal Investigator — Gustave Roussy center, Villejuif, France
Locations (12):
- Belgium (2):
  - Institut Bordet, Brussels
  - UZ Leuven, Leuven
- France (9):
  - CHU Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut de cancerologie de Montpellier, Montpellier
  - Institut de cancerologie de Lorraine, Nancy
  - Institut Curie, Paris
  - Institut Universitaire Cancer Toulouse - Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Royal Marsden Hospital, London, United Kingdom

REFERENCES:
- [Derived] Prat M, Le Naour A, Coulson K, Lemee F, Leray H, Jacquemin G, Rahabi MC, Lemaitre L, Authier H, Ferron G, Barret JM, Martinez A, Ayyoub M, Delord JP, Gladieff L, Tabah-Fisch I, Prost JF, Couderc B, Coste A. Circulating CD14high CD16low intermediate blood monocytes as a biomarker of ascites immune status and ovarian cancer progression. J Immunother Cancer. 2020 Jun;8(1):e000472. doi: 10.1136/jitc-2019-000472. PMID 32503947